CLINICAL TRIAL: NCT00847275
Title: Behaviour and Cognitive Evaluation for Dialysis Elderly Patients
Brief Title: Behaviour and Cognitive Evaluation for Dialysis Elderly Patients (BCDE)
Acronym: BCDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 06/12-K
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Renal Insufficiency
Keywords: Elderly patients; renal insufficiency; gerontologic evaluation
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): "Exclusive nephrology follow-up" arm
  Interventions: Other: Exclusive nephrology follow-up
- 2 (Experimental): "Geriatric follow-up" arm
  Interventions: Other: Geriatric follow-up

INTERVENTIONS:
Other: Exclusive nephrology follow-up — 250 patients will be included and randomized in the "exclusive nephrology follow-up" arm will continue their usual nephrology follow-up with consultations every 6 months during 3 years for dialysis patients or with consultations every 6 months before dialysis, 3 months after starting dialysis and every 6 months for a total duration of 3 years for non-dialysis patients. In addition to their nephrology consultations, patients will benefit from a geriatric evaluation with MMS, GDS and ADL scoring.
  Arms: 1
Other: Geriatric follow-up — 250 patients will be included and randomized in "geriatric follow-up" arm will continue their usual nephrology follow-up with consultations every 6 months during 3 years for dialysis patients or with consultations every 6 months before dialysis, 3 months after starting dialysis and every 6 months for a total duration of 3 years for non-dialysis patients. Patients randomized in the "geriatric follow-up" arm will also have more complete tests to evaluate cognitive functions (memory, language and movements), psychological functions (depression and anxiety) and dependency in activities of daily living. Other tests will allow evaluate vision, audition, mobility and nutritional status.
  Arms: 2

SUMMARY:
The trial is a multicenter, prospective, randomized, open study. A total of 500 elderly patients aged over 75 years with renal insufficiency stage 5 will be included in the study after signed informed consent. Patients will be randomized 1/1 in two arms : 250 patients in the "exclusive nephrology follow-up" arm will continue their usual follow-up; 250 patients in the "geriatric follow-up" arm will have both their usual nephrology follow-up and a geriatric follow-up.The aim of the study is to determine if a systematized gerontologist evaluation delay the occurrence of a composite primary endpoint : death, dementia, depression and severe dependency. The hypothesis is that the functional and vital prognosis of a patient with renal insufficiency depends not only on common and classical factors but also on cognitive and psychological functions and dependence, particularly in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged of 75 years old or more,
* Chronic kidney disease stage 5 defined by :
* either an estimated GFR (MDRD) ≤ 15ml/mn/1,73 m² in a non-dialysis patient whatever the duration of previous monitoring by the nephrologist("Pre-dialysis cohort"),
* or a dialysis treatment started for more than 3 months and less than one year, whatever the duration of pre-dialysis follow-up by the nephrologist("post-dialysis cohort"),
* Signed and dated informed consent.

Exclusion Criteria:

* Moderately severe to severe dementia (MMS ≤ 15),
* Major depression and/or GDS-15 > 10/15,
* Severe dependency (ADL < 3/6),
* Psychosis, mutism or aphasia,
* Malignancy or any pathology with life expectancy < one year,
* Ongoing specialized geriatric care

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-07; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
First outcome reached among: - death, - occurrence of a severe dementia (MMS < 10),- major depression detected by GDS-15 > 10/15 and confirmed by DSM-IV criteria,- severe dependency (ADL < 3/6). | 3 years

SECONDARY OUTCOMES:
Secondary outcomes are: - cognitive, psychic and autonomy scores,- cardiovascular morbidity and mortality,- biological follow-up of chronic kidney disease including haemoglobin level. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ESNAULT, Profesor, Study Chair — CHU NICE; Christian COMBE, Profesor, Study Chair — University Hospital, Bordeaux; Muriel RAINFRAY, Profesor, Study Chair — University Hospital, Bordeaux; Tugdual TANQUEREL, Doctor, Study Chair — CHU Brest; Armelle TILLY-GENTRIC, Profesor, Study Chair — CHU de Brest; Mokhtar AMRANDI, Doctor, Study Chair — CH Cholet; Jacques d'AVIGNEAU, Doctor, Study Chair — CH Cholet; Patrice DETEIX, Profesor, Study Chair — University Hospital, Clermont-Ferrand; Bruno LESOURD, Profesor, Study Chair — University Hospital, Clermont-Ferrand; Bernadette FALLER, Colmar, Study Chair — CHU Colmar; Nathalie SCHMITT, Doctor, Study Chair — CHU Colmar; Philippe ZAOUI, Profesor, Study Chair — University Hospital, Grenoble; Claire MILLET, Doctor, Study Chair — University Hospital, Grenoble; Jean-Noël OTTAVIOLI, Doctor, Study Chair — CHD La Roche sur Yon; Pierre LERMITE, Doctor, Study Chair — CHD La Roche sur Yon; Eric BOULANGER, Doctor, Study Chair — CHRU LILLE; François PUISIEUX, Profesor, Study Chair — CHRU LILLE; Jean-Claude ALDIGIER, Profesor, Study Chair — University Hospital, Limoges; Jean-Pierre CHARMES, Doctor, Study Chair — University Hospital, Limoges; Maurice LAVILLE, Profesor, Study Chair — Hospices Civils de Lyon; Brigitte COMTE, Doctor, Study Chair — Hospices Civils de Lyon; Michel LABEEUW, Profesor, Study Chair — Hospices Civils de Lyon; Marc BONNEFOY, Profesor, Study Chair — Hospices Civils de Lyon; Philippe BRUNET, Profesor, Study Chair — CHU Marseille; Sylvie BONIN-GUILLAUME, Doctor, Study Chair — CHU Marseille; Bernard CANAUD, Profesor, Study Chair — University Hospital, Montpellier; Claude JEANDEL, Profesor, Study Chair — University Hospital, Montpellier; Catherine DELCROIX, Doctor, Study Chair — Nantes University Hospital; Gilles BERRUT, Profesor, Study Chair — Nantes University Hospital; Patrice BROCKER, Profesor, Study Chair — CHU NICE; Bernard BRANGER, Doctor, Study Chair — CHU Nîmes; Benoît de WAZIERES, Profesor, Study Chair — CHU Nîmes; François VRTOVSNIK, Profesor, Study Chair — AP-HP (Hôpital Bichat); Fannie ONEN, Doctor, Study Chair — AP-HP (Hôpital Bichat); Dominique JOLY, Doctor, Study Chair — AP-HP (Hôpital Necker); Gilbert DERAY, Profesor, Study Chair — AP-HP (La Pitié-Salpétrière); Marc VERNY, Profesor, Study Chair — AP-HP (La Pitié-Salpétrière); Marc SOUID, Doctor, Study Chair — CH Poissy; Marie-Gabrielle CORD'HOMME, Doctor, Study Chair — CH Poissy; Véronique JOYEUX, Doctor, Study Chair — CHU Rennes; Gwenaëlle SOST, Doctor, Study Chair — CHU Rennes; Dominique BESNIER, Doctor, Study Chair — CH Saint-Nazaire; Philippe LEROUX, Doctor, Study Chair — CH Saint-Nazaire; Philippe NICOUD, Doctor, Study Chair — CH Sallanches; Serge PAYRAUD, Doctor, Study Chair — CH Sallanches; Bruno MOULIN, Profesor, Study Chair — CHU Strasbourg; Georges KALTENBACH, Profesor, Study Chair — CHU Strasbourg; Eric MICHEZ, Doctor, Study Chair — CH Vannes; Jean-Max GOLDFARB, Doctor, Study Chair — CH Vannes; Marie-Paule GUILLODO-HAMELET, Doctor, Study Chair — Dialysis center - Brest; Mohammed HADJ-ABDELKADER, Doctor, Study Chair — University Hospital, Clermont-Ferrand; Elodie CRETEL-DURAND, Doctor, Study Chair — CHU Marseille; Pierre JOUANNY, Profesor, Study Chair — CHU Rennes; Sylvie HILY, Doctor, Study Chair — CHU Saint-Nazaire
Locations (1):
- CHU de Nantes, Nantes, France